CLINICAL TRIAL: NCT07351708
Title: Development and Validation of a Post-operative Risk Of Local Recurrence Model Integrating Serology and Evalution (PROMISE) in Local Advanced Rectal Cancer Receiving Neoadjuvant Therapy: a Multicenter Study
Acronym: PROMISE model
Status: Completed | Type: Observational
Sponsor: Cai Zerong (Other)
Responsible Party: Sponsor-Investigator, Cai Zerong, Deputy Director of the Department, Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Other Study IDs: 2025ZSLYEC-724; No.82573589 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2010-01

CONDITIONS: Locally Advanced Rectal Cancer (LARC)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The pathological specimens before operation and the specimens after operation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LR patients: Local recurrence (LR) was defined as recurrent rectal cancer within the pelvic, including-but not limited to- lateral nodal recurrence, presacral recurrence, anastomotic recurrence, or perineal recurrence.
- non-LR patients: Local recurrence (LR) was defined as recurrent rectal cancer within the pelvic, including-but not limited to- lateral nodal recurrence, presacral recurrence, anastomotic recurrence, or perineal recurrence.

SUMMARY:
Local recurrence (LR) in locally advanced rectal cancer (LARC) correlated with poor survival and impaired quality of life. The aim of this study was to develop and validate machine learning (ML) models integrating clinicopathological features and inflammatory signature to predict LR in LARC patients undergoing neoadjuvant therapy followed by total mesorectal excision.

DETAILED DESCRIPTION:
To address the gap in accessible and integrative risk prediction, this study aimed to develop and validate an interpretable machine learning model for the early prediction of postoperative local recurrence in LARC patients using a multicenter cohort. We employed SHapley Additive exPlanations (SHAP) analysis to elucidate feature importance and provide clear interpretations for individual predictions, with the ultimate goal of evaluating the model's clinical utility in guiding personalized patient management-particularly by identifying high-risk patients in clinical practice and informing tailored follow-up and treatment strategies to improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed cT>=3 or cN+ stage rectal cancer by pelvic MRI or enhanced CT scan;
2. Pathological proved primary rectal adenocarcinoma;
3. Recieved full-cource radiation or more than 3 cycles of chemotherapy before surgery;
4. Recieved radical tumor resection by TME surgery.

Exclusion Criteria:

1. Diganosed with any distant metastasis disease or locally unresectable disease before neoadjuvant treatment or surgery;
2. Recieved local resection surgery (R2 resection) or postoperative pathology confirmed positive surgical margins (R1 resection);
3. Patients who died due to intra- or post-operative complications;
4. Patient who die or relapse within 30 days after surgery;
5. Patients who had a prior history of malignancy within 5 years before surgery;
6. Patients who were loss of follow-up or had inadequate clinical data.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eight hundred and sixty-nine patients (median [interquartile range] age, 57 [48, 64] years; 70% [611/869] male) with LARC between January 2010 and December 2022 in SYSU6H served as the training cohort, while 1446 patients with LARC between January 2010 and December 2022 in CHH (median age, 62 [54, 69]; 62% [902/1446] male) were served as the validation cohort.
Sampling Method: Non-Probability Sample
Enrollment: 2315 (Actual)
Dates: Start 2010-01-06 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Local recurrence | From date of randomization until the date of death from local recurrence, assessed up to 120 months
  Local recurrence (LR) was defined as recurrent rectal cancer within the pelvic, including-but not limited to- lateral nodal recurrence, presacral recurrence, anastomotic recurrence, or perineal recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Zerong Cai, MD, Study Director — Sixth Affiliated Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No
Please contact us by Email.